CLINICAL TRIAL: NCT06807190
Title: A Multi-centre, Prospective, Open Label, Non-interventional, Single-armed, 52 Weeks Post-marketing Study to Investigate Safety and Clinical Parameters of Awiqli Once Weekly in Patients With Diabetes Mellitus Under Real-world Clinical Practice Setting in Japan
Brief Title: General Use-results Surveillance With Awiqli in Patients With Diabetes Mellitus
Status: Recruiting | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1436-7680; U1111-1286-0463 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin icodec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Awiqli: Participants with diabetes mellitus will be treated with commercially available Awiqli according to routine clinical practice at the discretion of the treating physician.
  Interventions: Drug: Insulin Icodec

INTERVENTIONS:
Drug: Insulin Icodec — Participants will be treated with commercially available Awiqli according to routine clinical practice at the discretion of the treating physician.
  Other Names: Awiqli

SUMMARY:
The purpose of the study is to investigate the safety and effectiveness of Awiqli in participants with diabetes mellitus under real world clinical practice in Japan. Participants will get Awiqli as prescribed by the study doctor. The study will last for about 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available Awiqli has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.
* Male or female with no age limitation.
* Diagnosis of diabetes mellitus. There is no limitation for type of diabetes mellitus and prior treatment for diabetes mellitus.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Treatment with any investigational drug within 30 days prior to enrolment into the study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Contraindication described in Japanese package insert.
* Participants showing hypoglycaemic symptoms.
* Participants with a history of hypersensitivity to any ingredients of this drug.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises patients who are diagnosed with diabetes mellitus and who agree to be treated with Awiqli after consultation with their physician independently from the decision to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Reactions (ARs) | From baseline (week 0) to end of study (week 52)
  Measured as number of events.

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | From baseline (week 0) to end of study (week 52)
  Measured as number of events.
Number of Serious Adverse Events (SAEs) | From baseline (week 0) to end of study (week 52)
  Measured as number of events.
Number of Serious Adverse Reactions (SARs) | From baseline (week 0) to end of study (week 52)
  Measured as number of events.
Change in Glycosylated Haemoglobin (HbA1c) | From baseline (week 0) to end of study (week 52)
  Measured as percentage (%) point of HbA1c.
Change in Fasting Plasma Glucose (FPG) | From baseline (week 0) to end of study (week 52)
  Measured as milligrams per decilitre (mg/dL).
Change in Diabetes Therapy-Related Quality Of Life (DTR-QOL) | From baseline (week 0) to end of study (week 52)
  DTR-QOL is a Japanese questionnaire assessing the influence of diabetes treatment on the individual health related quality of life on 4 domains: "burden on social activities and daily activities", "anxiety and dissatisfaction with treatment", "hypoglycaemia" and "satisfaction with treatment". DTR-QOL contains 29 questions and the response scale is a 7-point scale (1: strongly agree to 7: strongly disagree). The score of each item will be reversed so that "7: strongly disagree" represents the highest/desirable QOL. The total score, after simple addition of the item scores, is converted to 0 to 100 (best-case response is 100; worst case response is 0).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (43):
- Japan (43):
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Japan
  - Jinnouchi Hospital_Internal Medicine, Kumamoto, Kumamoto, Japan
  - Miyachi Clinic, Aichi
  - Clinic Tosaki, Aichi
  - Uenishi Internal Medicine Clinic, Aichi
  - Ichinomiyanishi Hospital, Aichi
  - Ohisama Clinic_Aomori, Aomori
  - Kakizaki Tonyobyo Naika Clinic, Aomori
  - Chiba Central Medical Center, Chiba
  - Kimitsu Chuo Hospital_Diabetology and Endocrinology, Chiba
  - Soyokaze CardioVascular Medicine and Diabetes Care, Ehime
  - Clinic Masae Minami, Fukuoka
  - Ito Naika Clinic_Internal Medicine, Fukuoka
  - Takabe Diabetes Clinic, Hyogogoken
  - Kagayaki Diabetes and Endocrinology Clinic Sannomiya_Diabetes Internal Medicine, Hyōgo
  - Matsuda Diabetes Clinic, Hyōgo
  - Hyogo Prefectural Awaji Medical Center_Diabetes and Endocrinology, Hyōgo
  - Mitoyo General Hospital_Internal Medicine, Kagawa
  - Yokohama Rosai Hospital_Diabetes and Endocrinology, Kanagawa
  - H.E.C Science Clinic, Kanagawa
  - Kikuchi Naika Clinic_Kanagawa, Kanagawa
  - Hotaruno hakuyukai Medical Corporation of Japan, Kisarazu-shi, Chiba
  - Kyoto University Hospital, Kyoto-shi, Kyoto
  - MG Clinic, Mie
  - Kanno Naika_Internal Medicine, Mitaka-shi, Tokyo
  - Minamiminowa Clinic_Internal Medicine and Endocrinology and Metabolism, Nagano
  - Minagawa Clinic Internal Medicine, Niigata
  - Kitakamiekimae Naika Clinic, Numakunai
  - Osaka General Hospital of West Japan Railway Company_Diabetes and Metabolism, Osaka
  - Ogawa Clinic, Osaka
  - Matsuda Gastroenterology and Diabetes Clinic, Osaka
  - Okamoto Clinic for Diabetes and Endocrinology, Ōita
  - Imari Arita Kyoritsu Hospital_Internal Medicine, Saga
  - Yamane Hospital, Shimane
  - Kikuchi Medical Clinic, Shizuoka
  - Aoi Clinic_Diabetes and Internal Medicine, Tokyo
  - The Jikei University Hospital Dept of Diabetes, Metabolic, Tokyo
  - Matsuura Clinic, Tokyo
  - Mishuku Hospital, Tokyo
  - Tokyo Kyosai Hospital_Diabetes and Endocrinology, Tokyo
  - Kanto Central Hospital of the Mutual Aid Association of Public School Teachers_Diabetes and Endocrinology, Tokyo
  - Tamacenter Clinic Mirai, Tokyo
  - Honda Clinic_Internal Medicine, Tottori

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com